CLINICAL TRIAL: NCT03083769
Title: Functional Genetic Variants Affecting Tacrolimus Trough Levels and Side Effects in Chinese Renal Transplantation.
Status: Completed | Type: Observational
Sponsor: Southern Medical University, China (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); 181 Central Hospital of the Chinese PLA (Other)
Responsible Party: Principal Investigator, Liang Li, professor, Southern Medical University, China
Other Study IDs: NFEC-2016-176
Record Dates: First submitted 2017-03-08; First posted 2017-03-20 (Actual); Results first posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-10

CONDITIONS: Transplantation
Keywords: tacrolimus; genetic variants; side effects

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Human genomic DNA was extracted from leukocytes in patients' peripheral blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: The retrospective cohort consists of about 839 kidney transplant recipients from Nanfang Hospital. These patients used tacrolimus as immunosuppressive drug for preventing the rejection.The side effects (acute rejection, nephrotoxicity and neurotoxicity) will be recorded.
- Cohort 2: The retrospective cohort consists of about 663 kidney transplant recipients from Guilin No. 924 Hospital. These patients used tacrolimus as immunosuppressive drug for preventing the rejection.The side effects (acute rejection, nephrotoxicity and neurotoxicity) will be recorded.

SUMMARY:
The purpose of this study is to determine whether functional genetic variants can affect tacrolimus dose corrected trough levels and associate with the side effects in Chinese renal transplant recipients.

DETAILED DESCRIPTION:
Tacrolimus is an effective immunosuppressive drug widely used in solid organ transplantation to prevent rejection. It is characterized by a narrow therapeutic range and large inter- and intra- individual variability in its pharmacokinetics. Many factors are associated with the variability. Of these factors, genetic factor play an important role. Full understanding of this mechanism is important for the personalized use of tacrolimus and reducing the risk of side effects.The CYP3A5*3 (A6986G) resulting in a splicing defect and the absence of protein activity, was identified as a functional variant (Kuehl P.2001). The CYP3A4*1G was also reported as a functional variant (Richards-Waugh LL. 2014). In addition, other functional variants will also be identified and analyzed in our project.

Our project has two parts:first, retrospective study, 839 renal transplant recipients using tacrolimus as immunosuppressive drug were recruited from Nanfang Hospital. Fifty-eight SNPs from GWAS, GTEx and promoter region of CYP3A gene were genotyped. The association of 58 SNPs on the dose corrected tacrolimus trough levels and side effects (acute rejection, nephrotoxicity and neurotoxicity) were analyzed. Luciferase reporter gene assay were used to identify the functional variants. Second, in this part, there is another renal transplantation cohort. For this cohort, it was a retrospective cohort. All the patients will be stratified to different groups according to the different genotypes. The side effects (acute rejection, nephrotoxicity and neurotoxicity) will be observed.During the study period, all the therapeutic procedures of the patients are as usual.

This will be the largest cohort of this kind of study in Chinese population. The findings will be useful for the patients to improve the therapeutic efficacy and reduce the side effects.

ELIGIBILITY:
Inclusion Criteria:

Subject has been conducted kidney transplantation. Subject has used tacrolimus as immunosuppressant.

Exclusion Criteria:

Simultaneous liver-kidney transplantation. Patients with age less than 18 years old. Tacrolimus blood concentration monitoring less than 3 times. Failed to extract DNA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of the renal transplant recipients who received tacrolimus as immunosuppressant from Nanfang Hospital and Guilin No.924 Hospital. All the patients are Chinese.
Sampling Method: Probability Sample
Enrollment: 1502 (Actual)
Dates: Start 1998-01-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Nanfang Hospital, Guangzhou, Guangdong
  - Guilin No.924 Hospital, Guilin, Guangxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maseko N, Yang S, Li C, Zhang S, Wang R, Zhang Y, Li C, Zhang C, Li L. Impact of genetic polymorphisms on tacrolimus trough blood concentration in Chinese liver transplant recipients. Pharmacogenomics. 2023 Mar;24(4):207-217. doi: 10.2217/pgs-2022-0180. Epub 2023 Mar 17. PMID 36927114
- [Derived] Yang S, Jiang H, Li C, Lu H, Li C, Ye D, Qi H, Xu W, Bao X, Maseko N, Zhang S, Shao R, Li L. Genomewide association study identifies a novel variant associated with tacrolimus trough concentration in Chinese renal transplant recipients. Clin Transl Sci. 2022 Nov;15(11):2640-2651. doi: 10.1111/cts.13388. Epub 2022 Aug 28. PMID 35977080

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2
Started | 839 | 663
Completed | 819 | 631
Not Completed | 20 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Total
Number analyzed (Participants) | 839 | 663 | 1502
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.6) | 40.8 (10.6) | 41.1 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 263 | 189 | 452
  Male | 576 | 474 | 1050
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 839 | 663 | 1502
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 839 | 663 | 1502

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Rejection
Description: We will measure the number of participants with acute rejection during the day 1 to day 61 after transplantation. Kaplan-Meier analyses were performed for acute rejection in participants with different genotypes.
Time Frame: Day 1 to Day 61
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 819 | 631
participants | 256 | 37

2. Primary Outcome: Number of Participants With Tacrolimus-related Nephrotoxicities
Description: We will measure the number of participants with tacrolimus-related nephrotoxicities during the day 1 to day 61 after transplantation. Kaplan-Meier analyses were performed for tacrolimus-related nephrotoxicities in participants with different genotypes.
Time Frame: Day1 to Day 61
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 819 | 631
participants | 26 | 2

3. Primary Outcome: Number of Participants With Tacrolimus-related Neurotoxicities
Description: We will measure the number of participants with tacrolimus-related neurotoxicities during the day 1 to day 61 after transplantation. Kaplan-Meier analyses were performed for tacrolimus-related neurotoxicities in participants with different genotypes.
Time Frame: Day1 to Day 61
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2
Number analyzed (Participants) | 819 | 631
participants | 10 | 1

ADVERSE EVENTS:
Time Frame: Transplant recipients were followed for 61 days after transplantation to monitor side effects (acute rejection, nephrotoxicity and neurotoxicity).
Description: All the participants are at risk for All-Cause Mortality.
Arm/Group | Cohort 1 | Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/819 | 0/631
Serious Adverse Events (participants affected / at risk) | 256/819 | 37/631
Other Adverse Events (participants affected / at risk) | 0/819 | 0/631
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=819) | Cohort 2 (N=631)
Acute rejection (Renal and urinary disorders) | 256 (256) | 37 (37) — Acute rejection for kidney transplant recipients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-23): https://cdn.clinicaltrials.gov/large-docs/69/NCT03083769/Prot_SAP_000.pdf